CLINICAL TRIAL: NCT01212770
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Efficacy and Safety Study of Two Doses of Apremilast (CC-10004) in Subjects With Active Psoriatic Arthritis and a Qualifying Psoriasis Lesion
Brief Title: PALACE 3: Efficacy and Safety Study of Apremilast to Treat Active Psoriatic Arthritis
Acronym: PALACE 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-PSA-004
Record Dates: First submitted 2010-09-29; First posted 2010-10-01 (Estimated); Results first posted 2014-05-20 (Estimated); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; Psoriasis; Arthritis; inflammation; skin condition; inflammatory cells; apremilast; CC-10004; phosphodiesterase type 4
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis; Arthritis; Inflammation; Skin Diseases | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Apremilast 20 mg (Experimental): 20 mg Apremilast tablets administered twice daily for 24 weeks during the placebo-controlled phase followed by 20 mg Apremilast tablets administered twice daily for up to 4.5 years in the active treatment / long-term safety phase
  Interventions: Drug: Apremilast 20mg
- Apremilast 30 mg (Experimental): 30 mg Apremilast tablets administered twice a day for 24 weeks during the placebo-controlled phase followed by 30 mg Apremilast tablets administered twice a day for up to 4.5 years in the active treatment / long-term safety phase orally twice daily
  Interventions: Drug: Apremilast 30mg
- Placebo + 20 mg Apremilast (Placebo Comparator): Placebo + 20 mg Apremilast tablets administered twice daily for 24 weeks during the placebo-controlled phase followed by 20 mg Apremilast tablets administered twice daily for up to 4.5 years in the active treatment / long-term safety phase. Subjects who do not have at least 20% improvement in their swollen and tender joint counts at Week 16 will escape to 20 mg Apremilast twice daily at Week 16
  Interventions: Drug: Placebo
- Placebo + 30 mg Apremilast (Placebo Comparator): Placebo + 30 mg Apremilast tablets administered twice daily for 24 weeks during the placebo-controlled phase followed by 30 mg Apremilast tablets administered twice daily for up to 4.5 years in the active treatment / long-term safety phase. Subjects who do not have at least 20% improvement in their swollen and tender joint counts at Week 16 will escape to 30 mg Apremilast twice daily at Week 16.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apremilast 20mg — Apremilast 20 mg twice daily, orally
  Other Names: CC-10004
  Arms: Apremilast 20 mg
Drug: Apremilast 30mg — Apremilast 30 mg twice daily, orally
  Other Names: CC-10004
  Arms: Apremilast 30 mg
Drug: Placebo
  Arms: Placebo + 20 mg Apremilast; Placebo + 30 mg Apremilast

SUMMARY:
The purpose of this study is to determine whether apremilast is safe and effective in the treatment of patients with psoriatic arthritis and a qualifying psoriasis lesion.

Apremilast is proposed to improve signs and symptoms of psoriatic arthritis (tender and swollen joints, pain, physical function) in treated patients.

DETAILED DESCRIPTION:
Psoriatic arthritis (PsA) is an inflammatory arthritis that occurs in 6-39% of psoriasis patients. The immunopathogenesis of PsA, which mirrors but is not identical to that seen in psoriatic plaques, reflects a complex interaction among resident dendritic, fibroblastic and endothelial cells, and inflammatory cells attracted to the synovium by cytokines and chemokines. Apremilast (CC-10004) is a novel oral agent that modulates multiple inflammatory pathways through targeted phosphodiesterase type 4 (PDE4) enzyme inhibition. Therefore, apremilast has the potential to be effective in the treatment of PsA.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged ≥ 18 years at time of consent.
* Have a diagnosis of Psoriatic Arthritis (PsA, by any criteria) of ≥ 6 months duration.
* Meet the Classification Criteria for Psoriatic Arthritis (CASPAR) criteria for PsA at time of screening.
* Must have been inadequately treated by disease-modifying antirheumatic drugs (DMARDs)
* May not have axial involvement alone
* Concurrent Tx allowed with methotrexate, leflunomide, or sulfasalazine
* Have ≥ 3 swollen AND ≥ 3 tender joints.
* Males & Females must use contraception
* Stable dose of NSAIDs, narcotics and low dose oral corticosteroids allowed.
* Have at least one ≥2 cm psoriasis lesion

Exclusion Criteria:

* Pregnant or breast feeding.
* History of allergy to any component of the investigational product Hepatitis B surface antigen and/or Hepatitis C antibody positive at screening.
* Therapeutic failure on > 3 agents for PsA or > 1 biologic tumor necrosis factor (TNF) blocker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2010-09-30 (Actual); Primary Completion 2012-08-21 (Actual); Study Completion 2017-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (91):
- United States (23):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Catalina Pointe Clinical Research Incorporated, Tucson, Arizona
  - Bakersfield Dermatology and Skin Cancer Medical Group, Bakersfield, California
  - Dermatology Research Associates, Los Angeles, California
  - Desert Medical Advances, Palm Desert, California
  - Joao Nascimento, MD, Bridgeport, Connecticut
  - In Vivo Clinical Research, Doral, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Rheumatology Associates of Long Island, Orlando, Florida
  - Advent Clinical Research, Pinellas Park, Florida
  - Rockford Orthopedic Associates, LLC, Rockford, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - DermResearch, PLLC, Louisville, Kentucky
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - STAT Research, Inc., Dayton, Ohio
  - West Tennessee Research Institute, Jackson, Tennessee
  - Austin Dermatology Associates, Austin, Texas
  - Austin Regional Clinic, Austin, Texas
  - Center for Clinical Studies, Houston, Texas
  - Houston Medical Research, Houston, Texas
  - Texas Research Center, Sugar Land, Texas
- Australia (8):
  - Royal Prince Alfred Hospital, Camperdown
  - Skin Cancer Foundation, Carlton
  - Coff's Clinical Trials, Coffs Harbour
  - Heidelberg Repatriation Hospital, Heidelberg
  - Menzies Centre for Population Health Research, Hobart
  - Optimus Clinical Research Pty. Ltd, Kogarah
  - Coastal Joint Care, Maroochydore
  - The Queen Elizabeth Hospital, Woodville
- Canada (7):
  - Arthritis Research Centre of Canada, Vancouver, British Columbia
  - PerCuro Clinical Research, Victoria, British Columbia
  - Manitoba Clinic, Winnipeg, Manitoba
  - Arthritis Centre, Winnipeg, Manitoba
  - Alpha Clinical Research, LLC, St. John's, Newfoundland and Labrador
  - Niagara Peninsula Arthritis Centre Inc., St. Catharines, Ontario
  - Manna Research, Toronto, Ontario
- Finland (3):
  - Helsingin Reumakeskus Oy, Helsinki
  - Helsingin yliopistollinen keskussairaala, Helsinki
  - Finnish Medical Research Co, Pori
- France (4):
  - Centre Hospitalier Sud Francilien - Site Gilles de Corbeil, Corbeil-Essonnes
  - Hôtel-Dieu, Nantes
  - Groupe Hospitalier Archet I et II, Nice
  - Hopital Larrey Universite Paul Sabatier, Toulouse
- Germany (4):
  - Charite - Universitätsmedizin Berlin, Berlin
  - Klinische Forschung Berlin - Buch GmbH, Berlin
  - Klinikum der Friedrich-Schiller-Universität Jena, Jena
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
- Italy (2):
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico S.Orsola-Malpighi, Bologna
  - Fondazione PTV Policlinico Tor Vergata, Roma
- Lithuania (4):
  - Hospital of Lithuanian University Health and Sciences, Kaunas
  - Klaipeda University Hospital, Klaipėda
  - Panevezys Hospital, Panevezys
  - Siauliai Hospital, Šiauliai
- Poland (5):
  - Gabinet Internistyczno-Reumatologiczny Piotr Adrian Klimiuk, Bialystok
  - Centrum Medyczne Silesiana Sp. z o.o., Bytom
  - Malopolskie Centrum Medyczne S.C., Krakow
  - Prywatna Praktyka Lekarska Pawel Hrycaj, Poznan
  - REUMATIKA-Centrum Reumatologii Niepubliczny Zaklad Opieki Zdrowotnej, Warsaw
- Romania (6):
  - Baia Mare, Emergency County Hospital "Dr. Constantin Opris", Baia Mare
  - SC Duo Medical SRL, Bucharest
  - Sf. Maria Clinical Hospital, Bucharest
  - Emergency County Clinical Hospital, Cluj-Napoca
  - Sf Apostol Andrei Emergency Clinical County Hospital, Galati
  - C.M.I. Dr. Ciornohuz Adriana, Iași
- Russia (5):
  - Research Medical Complex Vashe Zdorovie, Kezch
  - Research Institute of Clinical and Experimental Lymphology, Novosibirsk
  - Penza Regional Clinical Hospital n.a. N.N. Burdenko, Penza
  - City Hospital 26, Saint Petersburg
  - Sverdlovsk Regional Clinical Hospital 1, Yekaterinburg
- Slovakia (3):
  - Narodny ustav reumatickych chorob, Piešťany
  - MUDr. Zuzana Cizmarikova, s.r.o., Poprad,Spisska Sobota
  - REUMEX s.r.o., Rimavská Sobota
- South Korea (7):
  - Hallym University Sacred Heart Hospital, Anyang, Kyunggi
  - Chungnam National University Hospital, Daejeon
  - Inha University Hosiptal, Incheon
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Ajou University Hospital, Suwon
- Spain (5):
  - Hospital Universitario a Coruna, A Coruña
  - Hospital de Basurto-Osakidetza, Bilbao
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Infanta Sofia, San Sebastián de los Reyes
- Switzerland (3):
  - HFR Fribourg - Hôpital Cantonal, Fribourg
  - Chuv Bh-04, Lausanne
  - Kantonsspital St. Gallen, Sankt Gallen
- United Kingdom (2):
  - Haywood Hospital, Burslem
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Result] Edwards CJ, Blanco FJ, Crowley J, Birbara CA, Jaworski J, Aelion J, Stevens RM, Vessey A, Zhan X, Bird P. Apremilast, an oral phosphodiesterase 4 inhibitor, in patients with psoriatic arthritis and current skin involvement: a phase III, randomised, controlled trial (PALACE 3). Ann Rheum Dis. 2016 Jun;75(6):1065-73. doi: 10.1136/annrheumdis-2015-207963. Epub 2016 Jan 20. PMID 26792812
- [Derived] Mease PJ, Hatemi G, Paris M, Cheng S, Maes P, Zhang W, Shi R, Flower A, Picard H, Stein Gold L. Apremilast Long-Term Safety Up to 5 Years from 15 Pooled Randomized, Placebo-Controlled Studies of Psoriasis, Psoriatic Arthritis, and Behcet's Syndrome. Am J Clin Dermatol. 2023 Sep;24(5):809-820. doi: 10.1007/s40257-023-00783-7. Epub 2023 Jun 14. PMID 37316690
- [Derived] Mease PJ, Gladman DD, Kavanaugh A, McGonagle D, Nash P, Guerette B, Nakasato P, Brunori M, Teng L, McInnes IB. Articular and Extra-Articular Benefits in ACR20 Non-responders at Week 104 Treated With Apremilast: Pooled Analysis of Three Randomized Controlled Trials. Rheumatol Ther. 2021 Dec;8(4):1677-1691. doi: 10.1007/s40744-021-00369-x. Epub 2021 Sep 18. PMID 34536218
- [Derived] Mease PJ, Gladman DD, Ogdie A, Coates LC, Behrens F, Kavanaugh A, McInnes I, Queiro R, Guerette B, Brunori M, Teng L, Smolen JS. Treatment-to-Target With Apremilast in Psoriatic Arthritis: The Probability of Achieving Targets and Comprehensive Control of Disease Manifestations. Arthritis Care Res (Hoboken). 2020 Jun;72(6):814-821. doi: 10.1002/acr.24134. Epub 2020 May 8. PMID 31909868
- [Derived] Kavanaugh A, Gladman DD, Edwards CJ, Schett G, Guerette B, Delev N, Teng L, Paris M, Mease PJ. Long-term experience with apremilast in patients with psoriatic arthritis: 5-year results from a PALACE 1-3 pooled analysis. Arthritis Res Ther. 2019 May 10;21(1):118. doi: 10.1186/s13075-019-1901-3. PMID 31077258
- [Derived] Gladman DD, Kavanaugh A, Gomez-Reino JJ, Wollenhaupt J, Cutolo M, Schett G, Lespessailles E, Guerette B, Delev N, Teng L, Edwards CJ, Birbara CA, Mease PJ. Therapeutic benefit of apremilast on enthesitis and dactylitis in patients with psoriatic arthritis: a pooled analysis of the PALACE 1-3 studies. RMD Open. 2018 Jun 27;4(1):e000669. doi: 10.1136/rmdopen-2018-000669. eCollection 2018. PMID 30018799

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 78 study centers in 16 countries.
Pre-assignment Details: This study consisted of a 24-week randomized, double-blind, placebo-controlled phase, a 28-week randomized, double-blind active treatment phase and a 4-year open-label safety phase, for an overall study duration of 5 years.
Groups:
- Placebo: Participants initially randomized to receive placebo tablets twice daily (BID) in the 24-week placebo-controlled phase. Participants who did not have at least 20% improvement in swollen and tender joint counts at Week 16 were re-randomized to either 20 mg or 30 mg apremilast twice daily (early escape).
- Apremilast 20 mg: Participants initially randomized to receive 20 mg apremilast tablets twice daily in the 24-week placebo-controlled phase continued receiving 20 mg apremilast tablets twice daily in the active treatment / long-term safety phase (LTSP).
- Apremilast 30 mg: Participants initially randomized to receive 30 mg apremilast tablets twice daily during the 24-week placebo-controlled phase continued receiving 30 mg apremilast tablets twice daily in the active treatment / long-term safety phase.
- Placebo / Apremilast 20 mg EE: Participants initially randomized to placebo twice daily were re-randomized due to early escape (EE) at Week 16 and began to receive 20 mg apremilast twice a day in the active treatment phase.
- Placebo / Apremilast 20 mg XO: Participants initially randomized to receive placebo twice daily were re-randomized at Week 24 (XO) to 20 mg apremilast tablets twice daily in the active treatment phase.
- Placebo / Apremilast 30 mg EE: Participants initially randomized to placebo twice daily were re-randomized due to early escape (EE) at Week 16 began receiving 30 mg apremilast tablets twice daily in the active treatment phase.
- Placebo / Apremilast 30 mg XO: Participants initially randomized to placebo twice daily were re-randomized at Week 24 to 30 mg apremilast twice daily in the active treatment phase.
- Placebo/Apremilast 20 mg (Long-Term Safety Phase): Participants initially randomized to placebo tablets twice daily during the 24-week placebo-controlled phase were re-randomized to 20 mg apremilast tablets twice daily at Week 16 or Week 24 and continued receiving apremilast 20 mg tablets twice daily in active treatment / long-term safety phase. (After 30 mg apremilast BID was identified as the optimal dose, all participants receiving 20 mg apremilast BID were switched to the 30 mg apremilast BID dose).
- Placebo/Apremilast 30 mg (Long-Term Safety Phase): Participants initially randomized to placebo tablets BID during the 24-week placebo-controlled phase were re-randomized to apremilast 30 mg tablets twice daily at Week 16 or Week 24 and continued receiving apremilast 30 mg tablets twice daily in the active treatment / long-term safety phase.
Period: Placebo-controlled Phase (Week 0 - 24)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo / Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg (Long-Term Safety Phase) | Placebo/Apremilast 30 mg (Long-Term Safety Phase)
Started | 169 | 169 | 167 | 0 | 0 | 0 | 0 | 0 | 0
Received Treatment | 169 | 169 | 167 | 0 | 0 | 0 | 0 | 0 | 0
Completed Week 16 | 156 | 157 | 156 | 0 | 0 | 0 | 0 | 0 | 0
Early Escape at Week 16 | 97 (1 participant who escaped early did not complete Week (Wk) 24) | 76 | 53 (1 participant who escaped early did not complete Week 24) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 146 | 147 | 145 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 23 | 22 | 22 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 10 | 12 | 8 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 6 | 5 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Miscellaneous | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Period: Active Treatment Phase (Weeks 25 - 52)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo / Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg (Long-Term Safety Phase) | Placebo/Apremilast 30 mg (Long-Term Safety Phase)
Started | 0 | 139 (8 participants who completed Week 24 did not enter the Week 24-52 active treatment phase) | 138 (7 participants who completed Week 24 did not enter the Week 24-52 active treatment phase) | 43 (3 participants who EE completed Week 24 did not enter the Week 24-52 active treatment phase) | 25 | 47 (3 participants who EE completed Week 24 did not enter the Week 24-52 active treatment phase) | 25 | 0 | 0
Completed | 0 | 120 | 126 | 32 | 23 | 44 | 23 | 0 | 0
Not Completed | 0 | 19 | 12 | 11 | 2 | 3 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 6 | 2 | 2 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 7 | 5 | 4 | 1 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 6 | 3 | 3 | 1 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Miscellaneous | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Period: Long-term Safety Phase (Year 2)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo / Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg (Long-Term Safety Phase) | Placebo/Apremilast 30 mg (Long-Term Safety Phase)
Started | 0 | 111 (9 participants who completed Week 52 did not enter the long-term safety phase (LTSP)) | 121 (5 participants who completed Week 52 did not enter the long-term safety phase) | 0 | 0 | 0 | 0 | 51 (Patients from the PBO/APR 20 mg EE and XO are combined;5 patients finished Wk 52;no entry into LTSP) | 64 (Patients from the PBO/APR 30 mg EE and XO are combined;3 patients finished Wk 52;no entry into LTSP)
Completed | 0 | 88 | 106 | 0 | 0 | 0 | 0 | 42 | 50
Not Completed | 0 | 23 | 15 | 0 | 0 | 0 | 0 | 9 | 14
Not completed — Adverse Event | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 6 | 7 | 0 | 0 | 0 | 0 | 4 | 6
Not completed — Non-compliance to study drug | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 9 | 3 | 0 | 0 | 0 | 0 | 4 | 4
Not completed — Lost to Follow-up | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Miscellaneous | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Period: Long-term Safety Phase (Year 3)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo / Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg (Long-Term Safety Phase) | Placebo/Apremilast 30 mg (Long-Term Safety Phase)
Started | 0 | 87 (1 participant who completed Year 2 did not continue treatment in Year 3) | 105 (1 participant who completed Year 2 did not continue treatment in Year 3) | 0 | 0 | 0 | 0 | 42 (The PBO/APR 20 mg EE and XO participants from week 24-52 are combined within the LTSP.) | 49 (Patients from the PBO/APR 30 mg EE and XO are combined;1 patient finished Wk 52;no entry into LTSP)
Completed | 0 | 76 (1 participant missed due to APR dispensed late) | 94 | 0 | 0 | 0 | 0 | 35 | 44
Not Completed | 0 | 11 | 11 | 0 | 0 | 0 | 0 | 7 | 5
Not completed — Adverse Event | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Lack of Efficacy | 0 | 3 | 4 | 0 | 0 | 0 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 3 | 4 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Miscellaneous | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Period: Long-term Safety Phase (Year 4)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo / Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg (Long-Term Safety Phase) | Placebo/Apremilast 30 mg (Long-Term Safety Phase)
Started | 0 | 77 (1 participant was counted in Year 4 but not in year 3 due to late APR dispensing) | 94 | 0 | 0 | 0 | 0 | 35 | 44
Completed | 0 | 71 | 83 | 0 | 0 | 0 | 0 | 32 | 42
Not Completed | 0 | 6 | 11 | 0 | 0 | 0 | 0 | 3 | 2
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 1 | 5 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Non-compliance with study drug | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Miscellaneous | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Long-term Safety Phase (Year 5)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo / Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg (Long-Term Safety Phase) | Placebo/Apremilast 30 mg (Long-Term Safety Phase)
Started | 0 | 70 (1 participant who completed Year 4 did not continue treatment in Year 5) | 83 | 0 | 0 | 0 | 0 | 32 | 42
Completed | 0 | 68 | 72 | 0 | 0 | 0 | 0 | 30 | 41
Not Completed | 0 | 2 | 11 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Missing | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Miscellaneous | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis dataset (FAS) consisted of all participants who were randomized as specified in the protocol.
Groups:
- Placebo: Participants initially randomized to receive placebo tablets twice daily.
- Apremilast 20 mg: Participants initially randomized to receive 20 mg apremilast tablets twice daily.
- Apremilast 30 mg: Participants initially randomized to receive 30 mg apremilast tablets twice daily.
- Total: Total of all reporting groups
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Total
Number analyzed (Participants) | 169 | 169 | 167 | 505
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (11.64) | 49.6 (12.10) | 49.9 (11.38) | 49.7 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 90 | 88 | 269
  Male | 78 | 79 | 79 | 236
Duration of psoriatic arthritis [Mean (Standard Deviation); unit: years] | 6.78 (6.463) | 7.74 (7.690) | 7.48 (7.646) | 7.33 (7.284)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 16
Description: Percentage of participants with an American College of Rheumatology 20% (ACR20) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 20% improvement in 78 tender joint count; • ≥ 20% improvement in 76 swollen joint count; and • ≥ 20% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); ◦ C-Reactive Protein.
Time Frame: Baseline and Week 16
Population: Full analysis set consisting of all participants randomized as specified in the protocol. Participants who withdrew early or who did not have sufficient data for a definitive determination of response status at Week 16 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 169 | 169 | 167
percentage of participants | 18.3 | 28.4 | 40.7
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; The percentage of participants with an ACR20 response was compared using a Cochran-Mantel- Haenszel (CMH) test. The Hochberg procedure was used to maintain the Type 1 error at the 0.05 significance level. The results were considered statistically significant if both the 30 mg apremilast dose versus placebo comparison and the 20 mg versus placebo comparison were statistically significant at the 0.05 significance level, or one of the comparisons was statistically significant at the 0.025 level; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted for baseline disease modifying antirheumatic drug (DMARD) use and and ≥ 3% body surface area (BSA) psoriasis involvement at baseline; Adjusted Difference = 22.3, 95% CI 2-sided [13.0 to 31.6] — Adjusted difference is the weighted average of the treatment differences across 4 strata of baseline DMARD use by ≥ 3% BSA psoriasis involvement at baseline with the CMH weights. The 95% CI is based on a normal approximation to the weighted average
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; In order to maintain the Type 1 error at the 0.05 significance level, the Hochberg procedure was to be used. The results of the endpoint were to be considered statistically significant if both the 30 mg apremilast dose versus placebo comparison and the 20 mg versus placebo comparison were statistically significant at the 0.05 significance level, or one of the comparisons was statistically significant at the 0.025 level; Test type: Superiority or Other; p = 0.0295, Cochran-Mantel-Haenszel; 2-sided p-value based on the Cochran-Mantel-Haenszel test adjusting for baseline DMARD use and ≥ 3% BSA psoriasis involvement at baseline; Adjusted Difference = 9.8, 95% CI 2-sided [1.1 to 18.6] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire- Disability Index (HAQ-DI) at Week 16
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire consisting of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and usual activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task are summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. Negative mean changes from Baseline in the overall score indicate improvement in functional ability.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline value and at least 1 postbaseline value at or prior to Week 16 are included; Last observation carried forward (LOCF) imputation was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 163 | 163 | 160
units on a scale | -0.065 (0.0335) | -0.131 (0.0337) | -0.192 (0.0339)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Pairwise comparisons (30 mg vs placebo and 20 mg vs placebo) were conducted conditional on the primary endpoint results. If the primary endpoint was statistically significant for both apremilast dose groups, pairwise comparisons for the HAQ-DI were to be evaluated at the 0.05 level using the Hochberg procedure. If only one apremilast dose was statistically significant, then only the comparison between that apremilast dose and placebo was conducted for the HAQ-DI score, at the 0.025 level; Test type: Superiority; p = 0.0073, ANCOVA; Based on an ANCOVA model with treatment group, baseline DMARD use and ≥ 3% BSA psoriasis involvement as factors and the baseline value as a covariate; LS Mean Difference = -0.127, 95% CI 2-sided [-0.220 to -0.034]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1619, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.066, 95% CI 2-sided [-0.158 to 0.027]

3. Secondary Outcome: Percentage of Participants With an ACR 20 Response at Week 24
Description: as for outcome 1
Time Frame: Baseline and Week 24
Population: Full analysis set; Participants who discontinued early, escaped early at Week 16 or who did not have sufficient data for a definitive determination of response status at Week 24 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 169 | 169 | 167
percentage of participants | 15.4 | 26.6 | 31.1
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0007, Cochran-Mantel-Haenszel — Secondary endpoints from the placebo-controlled period (Weeks 16 and 24) were analyzed in a hierarchical fashion to control the Type I error rate as described above; Two-sided p-value based on the Cochran-Mantel-Haenszel (CMH) test adjusting for baseline DMARD use and ≥ 3% BSA psoriasis involvement at baseline; Adjusted Difference = 15.5, 95% CI 2-sided [6.7 to 24.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.0110, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Adjusted Difference = 11.1, 95% CI 2-sided [2.7 to 19.5] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire- Disability Index (HAQ-DI) at Week 24
Description: as for outcome 2
Time Frame: Baseline and Week 24
Population: Full analysis set; participants with a baseline value and at least 1 postbaseline value at or prior to Week 24 are included; LOCF imputation was used. The Week 16 value was carried over to Week 24 for participants who escaped early at Week 16.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 163 | 164 | 161
units on a scale | -0.053 (0.0350) | -0.137 (0.0351) | -0.192 (0.0353)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Secondary endpoints from the placebo-controlled period (Weeks 16 and 24) were analyzed in a hierarchical fashion to control the Type I error rate as described above; Test type: Superiority; p = 0.0050, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.139, 95% CI 2-sided [-0.236 to -0.042]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0860, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.084, 95% CI 2-sided [-0.181 to 0.012]

5. Secondary Outcome: Change From Baseline in 36-item Short Form Health Survey (SF-36) Physical Functioning Domain at Week 16
Description: The Medical Outcome Study Short Form 36-Item Health Survey, Version 2 (SF-36) is a self-administered instrument that measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). Norm-based scores were used in analyses, calibrated so that 50 is the average score and the standard deviation equals 10. Higher scores indicate a higher level of functioning. The physical functioning domain assesses limitations in physical activities because of health problems. A positive change from Baseline score indicates an improvement.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline value and at least 1 postbaseline value at or prior to Week 16 are included; LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 162 | 162 | 160
units on a scale | 1.14 (0.589) | 2.29 (0.592) | 3.47 (0.594)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0053, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 2.32, 95% CI 2-sided [0.69 to 3.95]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.1658, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS mean Difference = 1.15, 95% CI 2-sided [-0.48 to 2.77]

6. Secondary Outcome: Percentage of Participants With a Modified Psoriatic Arthritis Response Criteria (PsARC) Response at Week 16
Description: Modified PsARC response is defined as improvement in at least 2 of the 4 measures, at least one of which must be tender joint count or swollen joint count, and no worsening in any of the 4 measures: • 78 tender joint count, • 76 swollen joint count, • Patient global assessment of disease activity, measured on a 100 mm visual Analog scale (VAS), where 0 mm = lowest disease activity and 100 mm = highest; • Physician global assessment of disease activity, measured on a 100 mm VAS, where 0 mm = lowest disease activity and 100 mm = highest. Improvement or worsening in joint counts is defined as decrease or increase, respectively, from baseline by ≥ 30%, and improvement or worsening in global assessments is defined as decrease or increase, respectively, from baseline by ≥ 20 mm VAS.
Time Frame: Baseline and Week 16
Population: Full analysis set; Participants who discontinued early, or who did not have sufficient data for a definitive determination of response status at Week 16 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 169 | 169 | 167
percentage of participants | 27.2 | 37.9 | 52.7
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Adjusted Difference = 25.4, 95% CI 2-sided [15.5 to 35.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0372, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Adjusted Difference = 10.4, 95% CI 2-sided [0.8 to 20.0] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Percentage of Participants Achieving a ≥ 75% Improvement in Psoriasis Area and Severity Index Score (PASI75) at Week 16
Description: The percentage of participants with Baseline psoriasis body surface area (BSA) involvement ≥ 3% who achieved 75% or greater improvement from Baseline in Psoriasis Area and Severity Index (PASI) score after 16 weeks of treatment. The Psoriasis Area and Severity Index (PASI) score is a combination of the intensity of psoriasis, assessed by erythema (reddening), induration (plaque thickness) and desquamation (scaling) scored on a scale from 0 (none) to 4 (very severe), together with the percentage of the area affected, rated on a scale from 0 (no involvement) to 6 (90% to 100% involvement). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline psoriasis involvement ≥ 3% of BSA are included; LOCF was used. Participants who did not have sufficient data (observed or imputed) for a determination of response status at Week 16 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 89 | 91 | 90
percentage of participants | 7.9 | 20.9 | 22.2
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0062, Cochran-Mantel-Haenszel; Two-sided p-value based on the Cochran-Mantel-Haenszel (CMH) test adjusting for baseline DMARD use; Adjusted Difference = 14.6, 95% CI 2-sided [4.5 to 24.8] — Adjusted difference is the weighted average of the treatment differences across 2 strata of baseline DMARD use with the CMH weights. The 95% CI is based on a normal approximation to the weighted average
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0134, Cochran-Mantel-Haenszel; Two-sided p-value based on the Cochran-Mantel-Haenszel (CMH) test adjusting for baseline DMARD use; Adjusted Difference = 13.0, 95% CI 2-sided [3.0 to 23.1] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain at Week 16
Description: The participant was asked to place a vertical line on a 100-mm visual analog scale on which the left-hand boundary (score = 0 mm) represents "no pain," and the right-hand boundary (score = 100 mm) represents "pain as severe as can be imagined." The distance from the mark to the left-hand boundary was recorded in millimeters.
Time Frame: Baseline and Week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 164 | 163 | 161
mm | -4.9 (1.79) | -8.6 (1.80) | -12.7 (1.81)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0021, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -7.8, 95% CI 2-sided [-12.8 to -2.9]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.1482, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -3.6, 95% CI 2-sided [-8.6 to 1.3]

9. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Entheses Score (MASES) at Week 16
Description: The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline MASES > 0 (i.e., pre-existing enthesopathy) and at least 1 postbaseline value at or prior to Week 16 are included; LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 106 | 93 | 107
units on a scale | -0.7 (0.27) | -0.7 (0.29) | -1.0 (0.27)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.5349, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-1.0 to 0.5]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.8231, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.7 to 0.9]

10. Secondary Outcome: Change From Baseline in Dactylitis Severity Score at Week 16
Description: Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present.
Time Frame: Baseline and Week 16
Population: Full analysis set. Participants with a baseline dactylitis severity score > 0 (i.e., pre-existing dactylitis) and at least 1 postbaseline value at or prior to Week 16 are included. LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 67 | 70 | 76
units on a scale | -1.3 (0.34) | -1.7 (0.33) | -2.1 (0.32)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0720, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.8, 95% CI 2-sided [-1.7 to 0.1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.3641, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.3 to 0.5]

11. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Week 16
Description: The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the: • 28 tender joint count (TJC), • 28 swollen joint count (SJC), • Patient's Global Assessment of Disease Activity measured on a 10 cm visual analog scale (VAS), where 0 cm = lowest disease activity and 10 cm = highest; • Physician's Global Assessment of Disease Activity -measured on a 10 cm VAS, where 0 cm = lowest disease activity and 10 cm = highest. The CDAI score ranges from 0-76 where lower scores indicate less disease activity. The following thresholds of disease activity have been defined for the CDAI: Remission: ≤ 2.8 Low Disease Activity: > 2.8 and ≤ 10 Moderate Disease Activity: > 10 and ≤ 22 High Disease Activity: > 22.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline value and at least 1 postbaseline value at or prior to Week 16 are included. LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 159 | 154 | 156
units on a scale | -2.76 (0.869) | -4.61 (0.886) | -7.70 (0.881)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -4.94, 95% CI 2-sided [-7.34 to -2.53]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.1325, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -1.85, 95% CI 2-sided [-4.27 to 0.56]

12. Secondary Outcome: Change From Baseline in the Disease Activity Score (DAS28) at Week 16
Description: The DAS28 measures the severity of disease at a specific time and is derived from the following variables: • 28 tender joint count • 28 swollen joint count, which do not include the distal interphalangeal (DIP) joints, the hip joint, or the joints below the knee; • C-reactive protein (CRP) • Patient's global assessment of disease activity. DAS28(CRP) scores range from 0 to approximately 10, with the upper bound dependent on the highest possible level of CRP. A DAS28 score higher than 5.1 indicates high disease activity, a DAS28 score less than 3.2 indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission.
Time Frame: Baseline and Week 16
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 163 | 160 | 160
units on a scale | -0.28 (0.084) | -0.54 (0.085) | -0.74 (0.085)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.47, 95% CI 2-sided [-0.70 to -0.24]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.0237, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.27, 95% CI 2-sided [-0.50 to -0.04]

13. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score at Week 16
Description: The FACIT-Fatigue scale is a 13-item self-administered questionnaire that assesses both the physical and functional consequences of fatigue. Each question is answered on a 5-point scale, where 0 means "not at all," and 4 means "very much." The FACIT-Fatigue scale score ranges from 0 to 52, with higher scores denoting lower levels of fatigue.
Time Frame: Baseline and Week 16
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 160 | 160 | 160
units on a scale | 1.18 (0.640) | 1.86 (0.643) | 3.72 (0.641)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0049, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 2.54, 95% CI 2-sided [0.77 to 4.30]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.4505, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 0.68, 95% CI 2-sided [-1.09 to 2.44]

14. Secondary Outcome: Change From Baseline in 36-item Short Form Health Survey (SF-36) Physical Functioning Domain at Week 24
Description: as for outcome 5
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Participants initially randomized to receive placebo tablets twice daily. Participants who did not have at least 20% improvement in swollen and tender joint counts at Week 16 were re-randomized to either to 20 mg or 30 mg apremilast twice daily (early escape).
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 162 | 163 | 161
units on a scale | 1.03 (0.581) | 2.71 (0.582) | 3.37 (0.585)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0043, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 2.34, 95% CI 2-sided [0.74 to 3.94]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.0404, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 1.67, 95% CI 2-sided [0.07 to 3.27]

15. Secondary Outcome: Percentage of Participants With a Modified Psoriatic Arthritis Response Criteria (PsARC) Response at Week 24
Description: as for outcome 6
Time Frame: Baseline and Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 169 | 169 | 167
percentage of participants | 23.1 | 32.0 | 44.3
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use and and involvement of >= 3% BSA with psoriasis at baseline; Adjusted Difference = 21.2, 95% CI 2-sided [11.5 to 30.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.0661, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use involvement of >= 3% BSA with psoriasis at baseline; Adjusted Difference = 8.7, 95% CI 2-sided [-0.5 to 18.0] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Percentage of Participants Achieving a ≥ 75% Improvement in Psoriasis Area and Severity Index Score (PASI75) at Week 24
Description: The percentage of participants with Baseline psoriasis body surface area (BSA) involvement ≥ 3% who achieved 75% or greater improvement from Baseline in Psoriasis Area and Severity Index (PASI) score after 24 weeks of treatment. The Psoriasis Area and Severity Index (PASI) score is a combination of the intensity of psoriasis, assessed by erythema (reddening), induration (plaque thickness) and desquamation (scaling) scored on a scale from 0 (none) to 4 (very severe), together with the percentage of the area affected, rated on a scale from 0 (no involvement) to 6 (90% to 100% involvement). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
Time Frame: Baseline and Week 24
Population: Full analysis set; participants with baseline psoriasis involvement ≥ 3% of BSA are included; LOCF was used. The Week 16 value was carried over to Week 24 for participants who escaped early. Participants who did not have sufficient data (observed or imputed) for a determination of response status at Week 24 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 89 | 91 | 90
percentage of participants | 11.2 | 22.2 | 25.6
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0099, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 14.8, 95% CI 2-sided [3.8 to 25.7] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.0515, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 10.8, 95% CI 2-sided [0.1 to 21.4] — [estimate comment as in outcome 7, analysis 1]

17. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain at Week 24
Description: as for outcome 8
Time Frame: Baseline and week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 164 | 164 | 162
mm | -4.4 (1.75) | -8.2 (1.76) | -10.9 (1.77)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0080, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS mean Difference = -6.6, 95% CI 2-sided [-11.4 to -1.7]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.1218, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -3.8, 95% CI 2-sided [-8.6 to 1.0]

18. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Entheses Score (MASES) at Week 24
Description: as for outcome 9
Time Frame: Baseline and week 24
Population: Full analysis set; participants with a baseline MASES > 0 (i.e., pre-existing enthesopathy) and at least 1 postbaseline value at or prior to Week 24 are included; LOCF imputation was used. The Week 16 value was carried over to Week 24 for participants who escaped early at Week 16.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 106 | 93 | 107
units on a scale | -0.7 (0.29) | -1.0 (0.31) | -1.1 (0.29)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.2761, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.3 to 0.4]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.5012, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-1.1 to 0.6]

19. Secondary Outcome: Change From Baseline in Dactylitis Severity Score at Week 24
Description: Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet will be rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present.
Time Frame: Baseline and Week 24
Population: Full analysis set. Participants with a baseline dactylitis severity score > 0 (i.e., pre-existing dactylitis) and at least 1 postbaseline value at or prior to Week 24 are included. LOCF was used. The Week 16 value was carried over to Week 24 for participants who escaped early at Week 16.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 67 | 71 | 77
units on a scale | -1.3 (0.35) | -1.7 (0.34) | -2.3 (0.32)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0399, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-1.9 to -0.0]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.4413, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.3 to 0.6]

20. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Week 24
Description: The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the: • 28 tender joint count (TJC), • 28 swollen joint count (SJC), • Patient's Global Assessment of Disease Activity measured on a 10 cm visual analog scale (VAS), where 0 cm = lowest disease activity and 10 cm = highest; • Physician's Global Assessment of Disease Activity -measured on a 10 cm VAS, where 0 cm = lowest disease activity and 10 cm = highest. The CDAI score ranges from 0-76 where lower scores indicate less disease activity. The following thresholds of disease activity have been defined for the CDAI: Remission: ≤ 2.8; Low Disease Activity: > 2.8 and ≤ 10; Moderate Disease Activity: > 10 and ≤ 22; High Disease Activity: > 22.
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 159 | 156 | 158
units on a scale | -2.53 (0.889) | -5.18 (0.900) | -7.81 (0.895)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -5.27, 95% CI 2-sided [-7.73 to -2.82]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.0349, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -2.65, 95% CI 2-sided [-5.11 to -0.19]

21. Secondary Outcome: Change From Baseline in the Disease Activity Score (DAS28) at Week 24
Description: The DAS28 measures the severity of disease at a specific time and is derived from the following variables: • 28 tender joint count • 28 swollen joint count, which do not include the DIP joints, the hip joint, or the joints below the knee; • C-reactive protein (CRP) • Patient's global assessment of disease activity. DAS28(CRP) scores range from 0 to approximately 10, with the upper bound dependent on the highest possible level of CRP. A DAS28 score higher than 5.1 indicates high disease activity, a DAS28 score less than 3.2 indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission.
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 163 | 161 | 161
units on a scale | -0.27 (0.087) | -0.57 (0.088) | -0.75 (0.087)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.48, 95% CI 2-sided [-0.72 to -0.24]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.0147, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.30, 95% CI 2-sided [-0.54 to -0.06]

22. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score at Week 24
Description: The FACIT-Fatigue scale is a 13-item self-administered questionnaire that assesses both the physical and functional consequences of fatigue. Each question is answered on a 5-point scale, where 0 means "not at all," and 4 means "very much." The FACIT-Fatigue scale score ranges from 0 to 52, with higher scores denoting lower levels of fatigue. A positive change from baseline score indicates an improvement.
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 161 | 163 | 161
units on a scale | 0.83 (0.652) | 2.01 (0.651) | 3.27 (0.654)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0078, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 2.44, 95% CI 2-sided [0.64 to 4.24]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.1936, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 1.19, 95% CI 2-sided [-0.61 to 2.98]

23. Secondary Outcome: Percentage of Participants With MASES Improvement ≥ 20% at Week 16
Description: Percentage of participants with pre-existing enthesopathy whose MASES improved by ≥ 20% from Baseline after 16 weeks of treatment. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline MASES > 0 (i.e., pre-existing enthesopathy) are included; LOCF was used. Participants who did not have sufficient data (observed or imputed) for a determination of response status at Week 16 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 109 | 97 | 112
percentage of participants | 53.2 | 48.5 | 54.5
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.7585, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use and involvement of >= 3% BSA with psoriasis at baseline; Adjusted Difference = 2.1, 95% CI 2-sided [-10.9 to 15.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.5808, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = -3.9, 95% CI 2-sided [-17.4 to 9.7] — [estimate comment as in outcome 1, analysis 1]

24. Secondary Outcome: Percentage of Participants With Dactylitis Improvement ≥ 1 Point at Week 16
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improved by ≥ 1 after 16 weeks of treatment. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline dactylitis severity score > 0 (i.e., pre-existing dactylitis) are included; LOCF was used. Participants who did not have sufficient data (observed or imputed) for a determination of response status at Week 16 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 71 | 71 | 80
percentage of participants | 59.2 | 66.2 | 71.3
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.1303, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD useinvolvement of >= 3% BSA with psoriasis at baseline; Adjusted Difference = 12.0, 95% CI 2-sided [-3.1 to 27.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.3610, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = 7.5, 95% CI 2-sided [-8.3 to 23.2] — [estimate comment as in outcome 1, analysis 1]

25. Secondary Outcome: Percentage of Participants With Good or Moderate European League Against Rheumatism (EULAR) Response at Week 16
Description: A EULAR response reflects an improvement in disease activity and an attainment of a lower degree of disease activity based on the DAS-28 score. A Good Response is defined as an improvement (decrease) in the DAS28 of more than 1.2 compared with Baseline and attainment of a DAS28 score less than or equal to 3.2. A Moderate Response is defined as either: • an improvement (decrease) in the DAS28 of greater than 0.6 and less than or equal to 1.2 and attainment of a DAS28 score of less than or equal to 5.1 or, • an improvement (decrease) in the DAS28 of more than 1.2 and attainment of a DAS28 score of greater than 3.2.
Time Frame: Baseline and Week 16
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 169 | 169 | 167
percentage of participants | 29.0 | 40.2 | 51.5
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = 22.5, 95% CI 2-sided [12.4 to 32.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.0309, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = 11.0, 95% CI 2-sided [1.2 to 20.9] — [estimate comment as in outcome 1, analysis 1]

26. Secondary Outcome: Percentage of Participants With MASES Improvement ≥ 20% at Week 24
Description: Percentage of participants with pre-existing enthesopathy whose MASES improved by ≥ 20% from Baseline after 24 weeks of treatment. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses.
Time Frame: Baseline and Week 24
Population: Full analysis set; participants with a baseline MASES > 0 are included; LOCF was used. The Week 16 value was carried over to Week 24 for participants who escaped early at Week 16. Participants who did not have sufficient data (observed or imputed) for a determination of response status at Week 24 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 109 | 97 | 112
percentage of participants | 51.4 | 51.5 | 54.5
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.5731, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = 3.8, 95% CI 2-sided [-9.1 to 16.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.8876, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = 1.0, 95% CI 2-sided [-12.6 to 14.6] — [estimate comment as in outcome 1, analysis 1]

27. Secondary Outcome: Percentage of Participants With Dactylitis Improvement ≥ 1 Point at Week 24
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improved by ≥ 1 after 24 weeks of treatment. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present.
Time Frame: Baseline and Week 24
Population: Full analysis set; participants with a baseline dactylitis severity score > 0 are included; LOCF was used. The Week 16 value was carried over to Week 24 for participants who escaped early at Week 16. Participants who did not have sufficient data (observed or imputed) for a determination of response status at Week 24 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 71 | 71 | 80
percentage of participants | 60.6 | 67.6 | 73.8
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.1172, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = 12.2, 95% CI 2-sided [-2.5 to 26.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.3695, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = 7.2, 95% CI 2-sided [-8.2 to 22.6] — [estimate comment as in outcome 1, analysis 1]

28. Secondary Outcome: Percentage of Participants With Good or Moderate EULAR Response at Week 24
Description: EULAR response reflects an improvement in disease activity and an attainment of a lower degree of disease activity based on the DAS-28 score. A Good Response is defined as an improvement (decrease) in the DAS28 of more than 1.2 compared with Baseline and attainment of a DAS28 score less than or equal to 3.2. A Moderate Response is defined as either: • an improvement (decrease) in the DAS28 of greater than 0.6 and less than or equal to 1.2 and attainment of a DAS28 score of less than or equal to 5.1 or, • an improvement (decrease) in the DAS28 of more than 1.2 and attainment of a DAS28 score of greater than 3.2.
Time Frame: Baseline and Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 169 | 169 | 167
percentage of participants | 20.1 | 32.0 | 42.5
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = 22.5, 95% CI 2-sided [13.0 to 32.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.0123, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = 11.7, 95% CI 2-sided [2.7 to 20.7] — [estimate comment as in outcome 1, analysis 1]

29. Secondary Outcome: Percentage of Participants With a ACR 50 Response at Week 16
Description: Percentage of participants with an American College of Rheumatology 50% (ACR50) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 50% improvement in 78 tender joint count; • ≥ 50% improvement in 76 swollen joint count; and • ≥ 50% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); ◦ C-Reactive Protein.
Time Frame: Baseline and Week 16
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 169 | 169 | 167
percentage of participants | 8.3 | 12.4 | 15.0
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0520, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = 6.8, 95% CI 2-sided [0.0 to 13.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.2052, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = 4.2, 95% CI 2-sided [-2.2 to 10.6] — [estimate comment as in outcome 1, analysis 1]

30. Secondary Outcome: Percentage of Participants With an ACR 70 Response at Week 16
Description: Percentage of participants with an American College of Rheumatology 70% (ACR70) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 70% improvement in 78 tender joint count; • ≥ 70% improvement in 76 swollen joint count; and • ≥ 70% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); ◦ C-Reactive Protein.
Time Frame: Baseline and Week 16
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 169 | 169 | 167
percentage of participants | 2.4 | 4.7 | 3.6
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.5154, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = 1.2, 95% CI 2-sided [-2.4 to 4.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.2527, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = 2.3, 95% CI 2-sided [-1.5 to 6.2] — [estimate comment as in outcome 1, analysis 1]

31. Secondary Outcome: Percentage of Participants With an ACR 50 Response at Week 24
Description: as for outcome 29
Time Frame: Baseline and Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 169 | 169 | 167
percentage of participants | 7.7 | 13.6 | 16.2
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0180, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = 8.3, 95% CI 2-sided [1.6 to 15.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.0807, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = 5.8, 95% CI 2-sided [-0.6 to 12.3] — [estimate comment as in outcome 1, analysis 1]

32. Secondary Outcome: Percentage of Participants With a ACR 70 Response at Week 24
Description: as for outcome 30
Time Frame: Baseline and Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 169 | 169 | 167
percentage of participants | 3.6 | 4.1 | 5.4
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.4230, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = 1.8, 95% CI 2-sided [-2.6 to 6.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.7870, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = 0.6, 95% CI 2-sided [-3.5 to 4.6] — [estimate comment as in outcome 1, analysis 1]

33. Secondary Outcome: Percentage of Participants Achieving a MASES Score of Zero at Week 16
Description: Percentage of participants with pre-existing enthesopathy whose MASES improves to 0 after 16 weeks of treatment. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses.
Time Frame: Week 16
Population: as for outcome 23
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 109 | 97 | 112
percentage of participants | 24.8 | 19.6 | 20.5
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.4707, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = -4.1, 95% CI 2-sided [-14.8 to 6.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.3547, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = -5.4, 95% CI 2-sided [-16.6 to 5.7] — [estimate comment as in outcome 1, analysis 1]

34. Secondary Outcome: Percentage of Participants Achieving a Dactylitis Score of Zero at Week 16
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improves to zero after 16 weeks of treatment. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present.
Time Frame: Week 16
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 71 | 71 | 80
percentage of participants | 35.2 | 40.8 | 41.3
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.4175, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = 6.6, 95% CI 2-sided [-8.6 to 21.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.4370, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = 6.4, 95% CI 2-sided [-9.1 to 21.8] — [estimate comment as in outcome 1, analysis 1]

35. Secondary Outcome: Percentage of Participants Achieving a MASES Score of Zero at Week 24
Description: Percentage of participants with pre-existing enthesopathy whose MASES improves to 0 after 24 weeks of treatment. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses.
Time Frame: Week 24
Population: as for outcome 26
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 109 | 97 | 112
percentage of participants | 28.4 | 20.6 | 27.7
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.9463, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = -0.4, 195% CI 2-sided [-12.1 to 11.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.2032, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = -7.7, 95% CI 2-sided [-19.3 to 3.8] — [estimate comment as in outcome 1, analysis 1]

36. Secondary Outcome: Percentage of Participants Achieving a Dactylitis Score of Zero at Week 24
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improves to zero after 24 weeks of treatment. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present.
Time Frame: Week 24
Population: as for outcome 27
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 71 | 71 | 80
percentage of participants | 36.6 | 45.1 | 46.3
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.2321, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = 9.8, 95% CI 2-sided [-5.8 to 25.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.2520, Cochran-Mantel-Haenszel; [statistical method as in outcome 15, analysis 2]; Adjusted Difference = 9.6, 95% CI 2-sided [-6.2 to 25.3] — [estimate comment as in outcome 1, analysis 1]

37. Secondary Outcome: Percentage of Participants With an ACR 20 Response at Week 52
Description: Percentage of participants with an American College of Rheumatology 20% (ACR20) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 20% improvement in 78 tender joint count; • ≥ 20% improvement in 76 swollen joint count; and • ≥ 20% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); ◦ C-Reactive Protein. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population consists of all participants who were randomized or re-randomized to apremilast at any time during the study. Only those participants who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo / Apremilast 20 mg: Participants who received placebo twice daily up to Week 16 or Week 24 and were then re-randomized to receive 20 mg apremilast twice daily.
- Placebo / Apremilast 30 mg: Participants who received placebo twice daily up to Week 16 or Week 24 and were then re-randomized to receive 30 mg apremilast twice daily.
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 54 | 67 | 116 | 127
percentage of participants | 59.3 [45.0 to 72.4] | 58.2 [45.5 to 70.2] | 56.0 [46.5 to 65.2] | 63.0 [54.0 to 71.4]

38. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) at Week 52
Description: as for outcome 2
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; participants with a Baseline value and a Week 52 value are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 55 | 67 | 122 | 127
units on a scale | -0.34 (0.407) | -0.34 (0.491) | -0.33 (0.505) | -0.35 (0.505)

39. Secondary Outcome: Change From Baseline in the SF-36 Physical Functioning Scale Score at Week 52
Description: as for outcome 5
Time Frame: Baseline and Week 52
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 55 | 66 | 121 | 127
units on a scale | 7.76 (8.236) | 6.87 (7.241) | 5.68 (8.467) | 5.87 (8.008)

40. Secondary Outcome: Percentage of Participants With a Modified PsARC Response at Week 52
Description: Modified PsARC response is defined as improvement in at least 2 of the 4 measures, at least one of which must be tender joint count or swollen joint count, and no worsening in any of the 4 measures: • 78 tender joint count, • 76 swollen joint count, • Patient global assessment of disease activity, measured on a 100 mm visual Analog scale (VAS), where 0 mm = lowest disease activity and 100 mm = highest; • Physician global assessment of disease activity, measured on a 100 mm VAS, where 0 mm = lowest disease activity and 100 mm = highest. Improvement or worsening in joint counts is defined as decrease or increase, respectively, from baseline by ≥ 30%, and improvement or worsening in global assessments is defined as decrease or increase, respectively, from baseline by ≥ 20 mm VAS. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; only those participants who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 53 | 66 | 116 | 124
percentage of participants | 81.1 [68.0 to 90.6] | 75.8 [63.6 to 85.5] | 71.6 [62.4 to 79.5] | 79.0 [70.8 to 85.8]

41. Secondary Outcome: Percentage of Participants Achieving a ≥ 75% Improvement in Psoriasis Area and Severity Index Score (PASI75) at Week 52
Description: The percentage of participants with Baseline psoriasis body surface area (BSA) involvement ≥ 3% who achieved 75% or greater improvement from Baseline in Psoriasis Area and Severity Index (PASI) score after 52 weeks. The Psoriasis Area and Severity Index (PASI) score is a combination of the intensity of psoriasis, assessed by erythema (reddening), induration (plaque thickness) and desquamation (scaling) scored on a scale from 0 (none) to 4 (very severe), together with the percentage of the area affected, rated on a scale from 0 (no involvement) to 6 (90% to 100% involvement). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; participants with Baseline Psoriasis Body Surface Area ≥ 3% and a Week 52 value are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 24 | 35 | 63 | 64
percentage of participants | 33.3 [15.6 to 55.3] | 28.6 [14.6 to 46.3] | 28.6 [17.9 to 41.3] | 39.1 [27.1 to 52.1]

42. Secondary Outcome: Change From Baseline in the Patient Assessment of Pain at Week 52
Description: as for outcome 8
Time Frame: Baseline and Week 52
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 55 | 66 | 122 | 127
mm | -19.9 (24.54) | -19.1 (26.95) | -14.9 (24.86) | -18.7 (27.01)

43. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Entheses Score (MASES) at Week 52
Description: as for outcome 9
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; participants with a baseline value > 0 (i.e., pre-existing enthesopathy) and a Week 52 value are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 34 | 48 | 66 | 87
units on a scale | -2.5 (3.10) | -2.2 (3.01) | -2.2 (2.98) | -1.9 (2.99)

44. Secondary Outcome: Change From Baseline in the Dactylitis Severity Score at Week 52
Description: as for outcome 19
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; participants with a baseline value > 0 (i.e., pre-existing dactylitis) and a Week 52 value are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 22 | 26 | 52 | 61
units on a scale | -3.1 (4.26) | -3.8 (4.52) | -2.9 (3.67) | -3.6 (4.30)

45. Secondary Outcome: Change From Baseline in the CDAI Score at Week 52
Description: The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the: •28 tender joint count (TJC), •28 swollen joint count (SJC), •Patient's Global Assessment of Disease Activity measured on a 10 cm visual analog scale (VAS), where 0 cm = lowest disease activity and 10 cm = highest; •Physician's Global Assessment of Disease Activity -measured on a 10 cm VAS, where 0 cm = lowest disease activity and 10 cm = highest. The CDAI score ranges from 0-76 where lower scores indicate less disease activity. The following thresholds of disease activity have been defined for the CDAI: Remission: ≤ 2.8 Low Disease Activity: > 2.8 and ≤ 10 Moderate Disease Activity: > 10 and ≤ 22 High Disease Activity: > 22.
Time Frame: Baseline and Week 52
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 53 | 66 | 116 | 124
units on a scale | -13.54 (10.689) | -12.38 (10.308) | -12.86 (12.654) | -14.14 (11.354)

46. Secondary Outcome: Change From Baseline in the DAS28 at Week 52
Description: The DAS28 measures the severity of disease at a specific time and is derived from the following variables: •28 tender joint count •28 swollen joint count, which do not include the DIP joints, the hip joint, or the joints below the knee; •C-reactive protein (CRP) •Patient's global assessment of disease activity. DAS28(CRP) scores range from 0 to approximately 10, with the upper bound dependent on the highest possible level of CRP. A DAS28 score higher than 5.1 indicates high disease activity, a DAS28 score less than 3.2 indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission.
Time Frame: Baseline and Week 52
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 54 | 67 | 121 | 127
units on a scale | -1.28 (1.102) | -1.29 (1.156) | -1.21 (1.063) | -1.41 (1.204)

47. Secondary Outcome: Change From Baseline in the FACIT-Fatigue Scale Score at Week 52
Description: as for outcome 22
Time Frame: Baseline and Week 52
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 54 | 65 | 121 | 127
units on a scale | 6.72 (8.996) | 5.66 (8.738) | 4.78 (8.526) | 6.20 (8.679)

48. Secondary Outcome: Percentage of Participants With MASES Improvement ≥ 20% at Week 52
Description: Percentage of participants with pre-existing enthesopathy whose MASES improved by ≥ 20% from Baseline after 52 weeks. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; participants with a baseline MASES > 0 (i.e., pre-existing enthesopathy) and who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 34 | 48 | 66 | 87
percentage of participants | 73.5 [55.6 to 87.1] | 75.0 [60.4 to 86.4] | 77.3 [65.3 to 86.7] | 71.3 [60.6 to 80.5]

49. Secondary Outcome: Percentage of Participants With Dactylitis Improvement ≥ 1 Point at Week 52
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improved by ≥ 1 after 52 weeks. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; Participants with a baseline dactylitis severity score > 0 (i.e., pre-existing dactylitis) and who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 22 | 26 | 52 | 61
percentage of participants | 95.5 [77.2 to 99.9] | 92.3 [74.9 to 99.1] | 88.5 [76.6 to 95.6] | 91.8 [81.9 to 97.3]

50. Secondary Outcome: Percentage of Participants Achieving Good or Moderate EULAR Response at Week 52
Description: A EULAR response reflects an improvement in disease activity and an attainment of a lower degree of disease activity based on the DAS-28 score. A Good Response is defined as an improvement (decrease) in the DAS28 of more than 1.2 compared with Baseline and attainment of a DAS28 score less than or equal to 3.2. A Moderate Response is defined as either: • an improvement (decrease) in the DAS28 of greater than 0.6 and less than or equal to 1.2 and attainment of a DAS28 score of less than or equal to 5.1 or, • an improvement (decrease) in the DAS28 of more than 1.2 and attainment of a DAS28 score of greater than 3.2. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: as for outcome 40
Measure: Number; unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 54 | 67 | 121 | 127
percentage of participants | 64.8 | 73.1 | 69.4 | 74.8

51. Secondary Outcome: Percentage of Participants With an ACR 50 Response at Week 52
Description: Percentage of participants with an American College of Rheumatology 50% (ACR50) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 50% improvement in 78 tender joint count; • ≥ 50% improvement in 76 swollen joint count; and • ≥ 50% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); ◦ C-Reactive Protein. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: as for outcome 40
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 53 | 66 | 119 | 126
percentage of participants | 28.3 [16.8 to 42.3] | 31.8 [20.9 to 44.4] | 25.2 [17.7 to 34.0] | 30.2 [22.3 to 39.0]

52. Secondary Outcome: Percentage of Participants With an ACR 70 Response at Week 52
Description: Percentage of participants with an American College of Rheumatology 70% (ACR70) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 70% improvement in 78 tender joint count; • ≥ 70% improvement in 76 swollen joint count; and • ≥ 70% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); ◦ C-Reactive Protein. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: as for outcome 40
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 53 | 67 | 120 | 125
percentage of participants | 20.8 [10.8 to 34.1] | 14.9 [7.4 to 25.7] | 9.2 [4.7 to 15.8] | 10.4 [5.7 to 17.1]

53. Secondary Outcome: Percentage of Participants Achieving a MASES Score of Zero at Week 52
Description: Percentage of participants with pre-existing enthesopathy whose MASES improves to 0 after 24 weeks. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; only those participants with a baseline value > 0 (i.e., pre-existing enthesopathy) and who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 34 | 48 | 66 | 87
percentage of participants | 44.1 [27.2 to 62.1] | 43.8 [29.5 to 58.8] | 33.3 [22.2 to 46.0] | 36.8 [26.7 to 47.8]

54. Secondary Outcome: Percentage of Participants Achieving a Dactylitis Score of Zero at Week 52
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improves to zero after 52 weeks. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Week 52
Population: as for outcome 49
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 22 | 26 | 52 | 61
percentage of participants | 68.2 [45.1 to 86.1] | 80.8 [60.6 to 93.4] | 75.0 [61.1 to 86.0] | 68.9 [55.7 to 80.1]

55. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) During the Placebo-Controlled Phase
Description: A TEAE is an adverse event (AE) with a start date on or after the date of the first dose of investigational product (IP) and no later than 28 days after the last dose of IP. An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. A serious AE is any AE that results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or constitutes an important medical event. For both AEs and SAEs the investigator assessed the severity of the event according to the grading scale: Mild: asymptomatic or with mild symptoms, Moderate: symptoms causing moderate discomfort or Severe: symptoms causing severe discomfort or pain.
Time Frame: Week 0 to Week 16 for placebo participants who entered EE at Week 16 and up to Week 24 for all other participants (placebo participants who remained on placebo through week 24 and participants randomized to the APR 20 mg BID or APR 30 mg BID)
Population: Safety population = participants who received at least one dose of IP;1 participant randomized to 30 mg APR who received PBO in error is counted in the PBO group;1 participant randomized to PBO who received 30 mg APR in error is counted in the 30 mg group;1 participant randomized to PBO who received 20 mg APR in error is counted in the 20 mg group
Measure: Number; unit: participants
Groups:
- Placebo: Participants received placebo tablets twice daily in the 24-week placebo-controlled phase. Participants who did not have at least 20% improvement in swollen and tender joint counts at Week 16 were rerandomized to either 20 mg or 30 mg apremilast twice daily (early escape).
- Apremilast 20 mg: Participants who received 20 mg apremilast tablets twice daily in the 24-week placebo-controlled phase.
- Apremilast 30 mg: Participants who received 30 mg apremilast tablets twice daily in the 24-week placebo-controlled phase.
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 168 | 170 | 167
participants
  Any TEAE | 83 | 100 | 104
  Any Drug-Related TEAE | 33 | 50 | 62
  Any Severe TEAE | 8 | 5 | 10
  Any Serious TEAE (SAE) | 9 | 3 | 6
  Any Serious Drug-Related TEAE | 2 | 0 | 0
  Any TEAE Leading to Drug Interruption | 4 | 20 | 16
  Any TEAE Leading to Drug Withdrawal | 10 | 13 | 12
  Any TEAE Leading to Death | 0 | 0 | 0

56. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events During the Apremilast Exposure Period
Description: as for outcome 55
Time Frame: Week 0 to Week 260; median duration of exposure to apremilast 20 mg BID was 121.71 weeks and 232.50 weeks for apremilast 30 mg BID
Population: Apremilast Subjects as Treated (AAT) were those who received at least 1 dose of apremilast at any time during the study. Participants were included in the treatment group corresponding to the apremilast dosing regimen they actually received, irrespective of the treatment group to which they were randomized or re-randomized.
Measure: Number; unit: participants
Groups:
- Apremilast 20 mg (Pre-switch): Participants who received apremilast 20 mg twice daily regardless of when the apremilast exposure started (at Week 0, 16, or 24). Only the TEAEs that occurred during apremilast 20 mg BID were counted.
- Apremilast 20/30 mg (Post-switch): Participants who switched from apremilast 20 mg BID to apremilast 30 mg BID. Only the TEAEs that occurred during APR 30 mg BID treatment were included.
- Apremilast 30 mg: Participants who received apremilast 30 mg twice daily regardless of when the apremilast-exposure started (at Week 0, 16, or 24).
Arm/Group | Apremilast 20 mg (Pre-switch) | Apremilast 20/30 mg (Post-switch) | Apremilast 30 mg
Number analyzed (Participants) | 241 | 97 | 242
participants
  Any TEAE | 194 | 64 | 209
  Any Drug-Related TEAE | 98 | 11 | 111
  Any Severe TEAE | 21 | 0 | 30
  Any Serious TEAE (SAE) | 38 | 4 | 54
  Any Serious Drug-Related TEAE | 5 | 0 | 3
  Any TEAE Leading to Drug Interruption | 48 | 4 | 53
  Any TEAE Leading to Drug Withdrawal | 30 | 0 | 30
  Any TEAE Leading to death | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: AEs are reported for the placebo-controlled phase from Week 0 to Week 16 for placebo participants who entered EE at Week 16 and up to Week 24 for all other participants and reported for the Apremilast Exposure Period from Week 0 to Week 260; median duration of apremilast 20 mg BID was 121.71 weeks and 232.50 weeks for apremilast 30 mg twice daily
Description: One participant randomized to 30 mg apremilast who received placebo in error is counted in the placebo group; one participant randomized to placebo who received 30 mg apremilast in error is counted in the 30 mg group; one participant randomized to placebo who received 20 mg apremilast in error is counted in the 20 mg group for safety analyses.
Groups:
- Weeks 0-24: Placebo (Placebo-Controlled Phase): Participants received placebo tablets twice daily during the placebo-controlled phase. Includes data through Week 16 for participants who escaped early, and through Week 24 for all other participants.
- Weeks 0-24: Apremilast 20 mg (Placebo- Controlled Phase): Participants received 20 mg apremilast tablets PO twice daily during the 24-week placebo-controlled phase.
- Weeks 0-24: Apremilast 30 mg (Placebo- Controlled Phase): Participants received 30 mg apremilast tablets PO twice daily during the 24-week placebo-controlled phase.
- APR Exposure Period Up to 5 Years: Apremilast 20 mg: Participants who received apremilast 20 mg twice daily regardless of when the apremilast exposure started (at Week 0, 16 or 24). Only TEAEs that occurred during apremilast 20 mg BID treatment (before the switch to 30 mg apremilast) were included.
- APR Exposure Period Up to 5 Years: Apremilast 20mg/30 mg: Participants who switched from apremilast 20 mg twice daily to apremilast 30 mg BID. Only the TEAEs that occurred during apremilast 30 mg twice daily treatment were included.
- APR Exposure Period Up to 5 Years: Apremilast 30 mg: Participants who received apremilast 30 mg twice daily throughout the study regardless of when the apremilast-exposure started (at Week 0, 16, or 24).
Arm/Group | Weeks 0-24: Placebo (Placebo-Controlled Phase) | Weeks 0-24: Apremilast 20 mg (Placebo- Controlled Phase) | Weeks 0-24: Apremilast 30 mg (Placebo- Controlled Phase) | APR Exposure Period Up to 5 Years: Apremilast 20 mg | APR Exposure Period Up to 5 Years: Apremilast 20mg/30 mg | APR Exposure Period Up to 5 Years: Apremilast 30 mg
Serious Adverse Events (participants affected / at risk) | 9/168 | 4/170 | 6/167 | 38/241 | 4/97 | 54/242
Other Adverse Events (participants affected / at risk) | 35/168 | 66/170 | 71/167 | 142/241 | 36/97 | 164/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Weeks 0-24: Placebo (Placebo-Controlled Phase) (N=168) | Weeks 0-24: Apremilast 20 mg (Placebo- Controlled Phase) (N=170) | Weeks 0-24: Apremilast 30 mg (Placebo- Controlled Phase) (N=167) | APR Exposure Period Up to 5 Years: Apremilast 20 mg (N=241) | APR Exposure Period Up to 5 Years: Apremilast 20mg/30 mg (N=97) | APR Exposure Period Up to 5 Years: Apremilast 30 mg (N=242)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary arteriovenous fistula (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acromegaly (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Intestinal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 1 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Toxic shock syndrome (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Cerebral haemorrhage traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Snake bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Whiplash injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Finger deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 2
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 2 | 0 | 7
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 1
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 2 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Breast enlargement (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ovarian haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Alcohol rehabilitation (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Weeks 0-24: Placebo (Placebo-Controlled Phase) (N=168) | Weeks 0-24: Apremilast 20 mg (Placebo- Controlled Phase) (N=170) | Weeks 0-24: Apremilast 30 mg (Placebo- Controlled Phase) (N=167) | APR Exposure Period Up to 5 Years: Apremilast 20 mg (N=241) | APR Exposure Period Up to 5 Years: Apremilast 20mg/30 mg (N=97) | APR Exposure Period Up to 5 Years: Apremilast 30 mg (N=242)
Diarrhoea (Gastrointestinal disorders) | 3 | 26 | 26 | 40 | 1 | 44
Nausea (Gastrointestinal disorders) | 9 | 19 | 23 | 28 | 3 | 47
Vomiting (Gastrointestinal disorders) | 1 | 5 | 8 | 10 | 1 | 14
Fatigue (General disorders) | 2 | 3 | 8 | 6 | 1 | 16
Bronchitis (Infections and infestations) | 2 | 3 | 1 | 17 | 3 | 20
Nasopharyngitis (Infections and infestations) | 2 | 7 | 4 | 34 | 12 | 36
Pharyngitis (Infections and infestations) | 1 | 1 | 1 | 14 | 1 | 14
Sinusitis (Infections and infestations) | 3 | 4 | 4 | 12 | 1 | 18
Upper respiratory tract infection (Infections and infestations) | 3 | 11 | 12 | 34 | 6 | 36
Urinary tract infection (Infections and infestations) | 1 | 2 | 5 | 19 | 3 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 4 | 9 | 0 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 12 | 4 | 18
Headache (Nervous system disorders) | 8 | 16 | 20 | 30 | 4 | 39
Insomnia (Psychiatric disorders) | 4 | 1 | 2 | 2 | 0 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 5 | 6 | 1 | 18
Hypertension (Vascular disorders) | 5 | 3 | 4 | 17 | 3 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications.